CLINICAL TRIAL: NCT03081988
Title: Prediction Model of Response for Combined Chemo-Radio-therapy Based on Clinical and Molecular Biology
Brief Title: Prediction Model of Response for CCRT in Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Su Youn Nam, Professor, Kyungpook National University Hospital
Other Study IDs: 2015R1D1A1A01059219
Record Dates: First submitted 2017-02-18; First posted 2017-03-17 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; chemoradiotherapy response; molecular factors
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — esophageal cancer tissue and paired normal tissue serum, plasma, buffy coat (DNA), whole blood (RNA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responder: Complete Remission after chemoradiotherapy in locally advanced or advanced esophageal cancer
  evaluation of disease status: endoscopy, CT, and/or PET-CT
  Interventions: Other: chemoradiotherapy
- non-responder: Progressive disease or stationary state after chemoradiotherapy in locally advanced or advanced esophageal cancer
  evaluation of disease status: endoscopy, CT, and/or PET-CT
  Interventions: Other: chemoradiotherapy

INTERVENTIONS:
Other: chemoradiotherapy — concomitant chemoradiotherpay is routine treatment in locally advanced and advanced esophageal cancer and it is not for research.

SUMMARY:
1. Retrospective review of old patients

   * Analysis of prediction factors for concomitant chemo-radiotherapy in locally advanced and advanced esophageal cancer from 2005 to 2015
2. Prospective case-control study: RNA sequencing & miRNA microarray

   * naive esophageal cancer patients who have a plan to receive concomitant chemo-radiotherapy

     * acquirement of tissue, blood, clinical information
     * isolation of RNA, DNA, serum database of clinical & demographic information

   ***Analysis of mRNA sequencing / miRNA sequencing**** first analysis of RNA sequencing: bioinformatician second analysis of RNA sequencing: principle investigator
3. Experimental set for qPCR (esophageal tissue) study group
4. TMA for screened exon gene
5. validation set for qPCR (esophageal tissue)
6. follow-up of circulating miRNA in blood (baseline blood & post-CCRT blood 3M, 6M, 12M)
7. Prediction model for CCRT response in esophageal Cancer based on clinical and molecular factors
8. Validate the prediction model.

DETAILED DESCRIPTION:
1. Retrospective review of old patients

   * Analysis of prediction factors for concomitant chemo-radiotherapy in locally advanced and advanced esophageal cancer from 2005 to 2015

   Study Group
   1. non responder
   2. CR but recurrence
   3. CR and survival loner than 2 years
2. Prospective case-control study: RNA sequencing & miRNA microarray

   * naive esophageal cancer patients who have a plan to receive concomitant chemo-radiotherapy --> acquirement of tissue, blood, clinical information --> isolation of RNA, DNA, serum database of clinical & demographic information

study group

1. non-responder (N=14)
2. Complete Remission (N=14)

   For considering the drop rate, 2-fold screening

   ***Analysis of mRNA sequencing / miRNA sequencing**** first analysis of RNA sequencing: bioinformatician second analysis of RNA sequencing: principle investigator

   3) Experimental set for qPCR (esophageal tissue) study group
   1. non-responder (N=40)
   2. complete remission (N=40)

   4) TMA for screened exon gene

   5) validation set for qPCR (esophageal tissue) new esophageal cancer set
   1. non-responder (N=30)
   2. complete remission (N=30)

   6) follow-up of circulating miRNA in blood (baseline blood & post-CCRT blood 3M, 6M, 12M)

   7) Prediction model for CCRT response in esophageal Cancer based on clinical and molecular factors

   Test several combination models
   1. gene + gene combination,
   2. gene + clinical information combination,
   3. gene + gene + clinical information combination

   8) Validate the prediction model.

   9) primary organoid culture and prediction of chemoradiotherapy response

ELIGIBILITY:
Inclusion Criteria:

1. locally advanced or advanced esophageal cancer who want concomitant chemoradiotherapy
2. persons who assigned the written informed consents.

Exclusion Criteria:

1. persons who did't assign the informed consents
2. other organ cancer
3. heavy alcoholics

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: locally advanced or advanced esophageal cancer who want concomitant chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2015-10-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction model for CCRT response based on clinical and genetic molecular factors | up to 36 months
  prediction model for CCRT response based on clinical and genetic molecular factors in esophageal cancer

SECONDARY OUTCOMES:
banking of remained human material for post genetic & molecular study | up to 10 years
  banking of remained human material for post genetic & molecular study
circulating preditction marker for CCRT response and prognosis | up to 5 years
  circulating miRNA sequencing
tissue prediction marker for CCRT response and prognosis | up to 5 years
  tissue RNA sequencing / tissue microarray
in-vitro prediction of CCRT using primary esophageal cancer organoid | up to 6 month
  1. Esophageal cancer derived primary organoid culture
  2. treat RT and 5-FU to esophageal cancer organoid
  3. measure the response of CCRT (live cell/dead cell)
     * This process is in-vitro process, not in-vivo experiment.

OTHER OUTCOMES:
Clinical prediction factors for CCRT response (retrospective study) | up to 5 years
  Evaluation of clinical prediction factors for CCRT response in esophageal cancer from 2005-2015 (retrospective study)

CONTACTS AND LOCATIONS:
Overall Officials: Su Youn Nam, MD, PhD, Principal Investigator — Kyungpook National University Medical Center
Locations (1):
- Kyungpook National University Medical Canter, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided